CLINICAL TRIAL: NCT04000113
Title: Therapeutic Effect of Laser Acupuncture on Insomnia in Perimenopausal Women : a Randomized, Double-blind Controlled Study
Brief Title: Therapeutic Effect of Laser Acupuncture on Insomnia in Perimenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Taipei Chinese Medical Association, Taiwan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-04-005C
Record Dates: First submitted 2019-05-19; First posted 2019-06-27 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Insomnia Type; Sleep Disorder; Perimenopausal Women
Keywords: menopause; insomnia; sleep disorder
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser acupuncture treatment (Experimental): Subjects accept low-dose near-infrared laser acupuncture (10mWx10) treatment for 5 minutes in each trial.
  Interventions: Device: laser acupuncture
- Sham laser acupuncture treatment (Sham Comparator): Subjects accept the sham (blank) laser acupuncture treatment for 5 minutes in each trial.
  Interventions: Device: Sham laser

INTERVENTIONS:
Device: laser acupuncture — low level laser emission on specific acupuncture points
  Arms: laser acupuncture treatment
Device: Sham laser — Sham laser
  Arms: Sham laser acupuncture treatment

SUMMARY:
According to previous studies, the quality of subjective sleep in women is generally worse than that of men. Although studies have shown that menopausal women who use hormone therapy can improve sleep disorders, the limited benefits of hormone therapy are reported, the duration of treatment and efficacy required is uncertain. The suspicions of the safety of hormone therapy have deterred many menopausal women.

Systematic review and meta-analysis show that acupuncture and related therapies (including electro-acupuncture, ear needle, body acupoint massage and ear acupoint massage, etc.) used in the study of insomnia treatment have a significant therapeutic effect. However, for the reason that most of them are invasive treatments, patients receiving such treatment are often afraid and hesitated. This study will apply the low-energy laser acupuncture treatment trials to menopausal women with insomnia. Sixty perimenopausal female volunteer subjects with 45-60 years of age who have been assessed and screened for sleep disorders will be recruited and participate in this experiment. After completing the basic data and various related scales, the subjects will undergo a double-blind, randomly allocated and controlled clinical trials. The experimental procedure is that the subjects will be placed in a soundproof, lying on a comfortable bed. After the instruments setting ready, subject receives the monitoring of 5-minute heart rate variability (HRV) measurements before and after the near-infrared laser acupuncture (10mWx10) treatment, a total of 30 minutes experimental process. The results of the analysis will be based on the Pittsburgh Sleep Quality index (PSQI) questionnaire, the Insomnia Severe Index scale (ISI) data as the main assessment results for analysis. The Menopause Rating Scale, (MRS), the Beck Depression Inventory Index scale (BDI-II) and the signal measurements of heart rate variability will be analyzed as secondary assessment grounds. Data of the questionnaires will be analyzed by the statistical method of Pair-t test for the comparison of the data before and after trial. The signal data of heart rate variability are analyzed by the two way ANOVA method. We expect that by way of combination of low-energy laser light irradiation method and theory of effective acupoints for insomnia can effectively improve the quality of sleep in peri-menopausal women.

DETAILED DESCRIPTION:
According to previous studies, the quality of subjective sleep in women is generally worse than that of men. The prevalence rate can be dramatically increased from 30% before menopause to 50% during menopausal transition. Although studies have shown that menopausal women who use hormone therapy can improve sleep disorders caused by hot flashes, night sweats, sleep disorders, such as sleep apnea, the limited benefits of hormone therapy are reported, the duration of treatment and efficacy required is uncertain. The doubts about the safety of hormone therapy have deterred many menopausal women.

Systematic review and meta-analysis show that acupuncture and related therapies (including electroacupuncture, ear needle, body acupoint massage and ear acupoint massage, etc.) used in the study of insomnia treatment have a significant therapeutic effect. However, for the reason that most of them are invasive treatments, patients receiving such treatment are often afraid and hesitated. This study will apply the low-energy laser acupuncture treatment trials to menopausal women with insomnia. Sixty perimenopausal female volunteer subjects with 45-60 years of age who have been assessed and screened for sleep disorders will be recruited and participate in this experiment. After completing the basic data and various related scales, the subjects will undergo a double-blind, randomly allocated and controlled clinical trials. The experimental procedure is that the subjects will be placed in a soundproof, undisturbed clinic room, lying on a comfortable bed and a pillow and covered by a thin blanket. After the instruments setting ready, subject lie by first for 10 minutes, then a 5-minute heart rate variability (HRV) measurement recording is underwent, followed by low-dose near-infrared laser acupuncture (10mWx10) treatment for 5 minutes, then subject lie by again for 5 minutes, and another 5 minutes of heart rate variability instrument recording followed, a total of 30 minutes experimental process. Acupoints of treatment will include both sides of the Sleep 1 (EXTRA-1), both sides of the Neiguan (PC-6), both sides of Shemen (HT-7), both sides of the Sanyinjiao (SP-3), both sides of the Taichung (LI-3),total of 10 acupoints. The results of the analysis will be based on the Pittsburgh Sleep Quality index (PSQI) questionnaire, the Insomnia Severe Index scale (ISI) data as the main assessment results for analysis. The Menopause Rating Scale, (MRS), the Beck Drepression Inventory Index scale (BDI-II) and the signal measurements of heart rate variability will be analyzed as secondary assessment grounds. Data of the questionnaires will be analyzed by the statistical method of Pair-t test for the comparison of the data before and after trial. The signal data of heart rate variability are analyzed by the two way ANOVA method. We expect that by way of combination of low-energy laser light irradiation method and theory of effective acupoint for insomnia can effectively improve the quality of sleep in perimenopausal women. The experiment will start on June, 2019.

ELIGIBILITY:
Inclusion Criteria:

* age of 45-60,irregular menstruation cycle at least 3 months or menopause for one year.
* clinical symptoms of insomnia attack 3times per-week for at least 3 months
* no hormone replacement therapy at least one month
* no problem on intellectual or text, verbal communication
* informed consent given

Exclusion Criteria:

* epilepsy, diabetic neuropathy,arrythmia, CAD, abnormal blood pressure, severe renal disease, several liver disease, endocrine or metabolic disease,malignant tumor disease, dermal diseae or cancer
* acute or infectious disease, fever.
* neurosensory or perception disturbance, inflammatory painful disease which affect sleep quality.
* depression, anxiety, schizophrenia or other psychological problem.
* parasomnia, obstructive sleep apnoea,rapid eye movement sleep disorder and restless legs syndrome.
* lifestyle without sleep routine
* hypnotics dependent for 6 months.
* any medicine or therapy for problem of menopause and autonomic nerve system in one month.
* photophobia
* drug, alcohol,caffeine abuse.
* attending any clinical trial for 3 months.
* coagulation disturbance

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — peri-menopausal transition
Enrollment: 60 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
the Pittsburgh Sleep Quality index (PSQI) questionnaire, | scores change between baseline and after last treatment(one month later)
  The 2I-item PSQI yields a global score, which represents the sum of seven individual component scores: sUbjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances (including items such as feeling pain, having difficulty breathing), use of medications for sleep and daytime dysfunction (including items related to daytime sleepiness and energy).
the Insomnia Severe Index scale (ISI) | scores change between baseline and after last treatment(two weeks and one month later)
  The Insomnia Severity Index (ISI) is composed of seven items that evaluate: (a) the severity of sleep-onset (initial), (b) sleep maintenance (middle), (c) early morning awakening (terminal) problems, (d) satisfaction with current sleep pattern, (e) interference with daily functioning, (f) noticeability of impairment attributed to the sleep problem, and (g) level of distress caused by the sleep problem. Each of these items is rated on a five-point Likert scale ("0" = not at all, "4"= extremely) and the time interval is "in the last 2 weeks". Total scores range from 0 to 28, with high scores indicating greater insomnia severity.

SECONDARY OUTCOMES:
The Menopause Rating Scale (MRS) | scores change between baseline and after last treatment(one month later)
  The score increases point by point with increasing severity of subjectively perceived symptoms in each of the 11 items (severity 0 [no complaints] 4 scoring points [very severe symptoms]). The respondent provides the subject's personal perception by checking one of 5 possible boxes of "severity" for each of the items.
The Beck Inventory Index scale (BDI-II) | scores change between baseline and after last treatment(one month later)
  The BDI-II is a 21-item self-report measure of the severity of depressive symptomatology. Each of the 21 items is rated on a 4-point scale ranging from 0-3. The rating are summed, yielding a total score that can range from 0-63.
The signal measurements of heart rate variability | change of nLF and HFcomponents of HRV from baseline and after last treatment.(one month later)
  Frequency-domain analysis of heart rate variability (HRV), a noninvasive method, has been used to reflect cardiac autonomic nervous activity in humans. The high-frequency power (HF; 0.15-0.4 Hz) of HRV represents vagal (parasympathetic) control of heart rate. The low-frequency power (LF; 0.04- 0.15 Hz) of HRV is jointly contributed by both sympathetic and vagal nerves, whereas normalized LF (nLF) is regarded as the sympathetic modulation.An elevated LF component and a decreased HF component of the HRV have been found in women with insomnia when they are compared with healthy women.

OTHER OUTCOMES:
sleep diary | scores change between baseline and after last treatment(one month later)
  The sleep diary provides daily subjective estimates of sleep parameters including: daytime nap, sleep aids intake, bedtime, sleep onset latency, frequency of nocturnal awakenings, awakenings duration, wake-up time, arising time, feeling upon arising (five-point scale) and sleep quality (five-point scale).

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Lin Yang, MD, PhD, Principal Investigator — Center for Traditional Medicine,Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No